CLINICAL TRIAL: NCT05918042
Title: Multicentre, Non-interventional, Observational, Prospective Study to Evaluate 1-st Line Treatment Approaches in HRD+ Ovarian Cancer Patients in Russian Federation
Brief Title: A Non-interventional Prospective Study of 1-st Line Treatment Approaches in OVArian Cancer Patients With HRD+ Status in Russian Federation
Acronym: OVARD
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133FR00195
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Study population will consist of HRD+ (BRCAm +/- positive genomic instability score according to used test system) OC with available medical history. It is estimated that approximately 400 patients will be enrolled in approximately 25 sites. Demographic and clinical characteristics, treatment approaches and outcomes in HRD+ patients with high-grade epithelial ovarian, primary peritoneal, and/or fallopian tube cancer will be collected at baseline and on prospective visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age;
* Willing and ability to provide written informed consent for participation in the study;
* Known status HRD+ (positive BRCAm test and/or positive Genomic Instability test);
* Patients with histologically confirmed diagnosis of high-grade IC-IV FIGO stages epithelial ovarian, primary peritoneal, and/or fallopian tube cancer;
* Completed primary treatment (surgery and/or 1st line CT +/- bevacizumab) no more than 3 months after completion of primary treatment.

Exclusion Criteria:

* Patients participating in other clinical studies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of HRD+ (BRCAm +/- positive genomic instability score according to used test system) OC with available medical history. It is estimated that approximately 400 patients will be enrolled in approximately 25 sites. Demographic and clinical characteristics, treatment approaches and outcomes in HRD+ patients with high-grade epithelial ovarian, primary peritoneal, and/or fallopian tube cancer will be collected at baseline and on prospective visits.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
To describe the demographic and clinical characteristics of the patient population with HRD-positive OC (HRD+ BRCAwt and HRD+ BRCAm) | 18 months
  Demographic and baseline clinical characteristics will be summarized descriptively for the entire cohort of eligible patients.

SECONDARY OUTCOMES:
To describe diagnostic and primary treatment approaches (surgery, first line chemotherapy+/-bevacizumab) of HRD+ with high-grade, epithelial ovarian, primary peritoneal, and/or fallopian tube cancer in routine practice | 18 months
  population and the maintenance regimens initiated after the primary OC therapy .
To describe first-line maintenance treatment approaches | 18 months
  population and the maintenance regimens initiated after the primary OC therapy .

CONTACTS AND LOCATIONS:
Locations (24):
- Russia (24):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Chelyabinsk
  - Research Site, Grozny
  - Research Site, Irkutsk
  - Research Site, Izhevsk
  - Research Site, Kaliningrad
  - Research Site, Kaluga
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Lyubertcy
  - Research Site, Moscow
  - Research Site, N.Novgorod
  - Research Site, Nal'chik
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Sochi
  - Research Site, Tomsk
  - Research Site, Ufa
  - Research Site, Vladivostok
  - Research Site, Yakutiya
  - Research Site, Yaroslavl